CLINICAL TRIAL: NCT05335447
Title: An Open-label Study in Healthy Male Subjects to Investigate the Metabolism and Excretion Pathways of GLPG3667 Following a Single Oral Dose of [14C]-GLPG3667 and to Determine the Absolute Bioavailability Relative to an Intravenous [14C]-GLPG3667 Microtracer
Brief Title: Evaluation of Mass Balance and Absolute Bioavailability of GLPG3667
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG3667-CL-107; 2021-006730-39 (EudraCT Number)
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1 - Absolute Bioavailability (Experimental)
  Interventions: Drug: GLPG3667 capsule; Drug: [14C]-GLPG3667 solution for infusion
- Period 2 - Mass Balance (Experimental)
  Interventions: Drug: [14C]-GLPG3667 capsule

INTERVENTIONS:
Drug: GLPG3667 capsule — On Day 1, participants will receive a single oral dose of GLPG3667
  Arms: Period 1 - Absolute Bioavailability
Drug: [14C]-GLPG3667 solution for infusion — On Day 1, participants will receive a single microtracer microdose of [14C]-GLPG3667 as an intravenous infusion
  Arms: Period 1 - Absolute Bioavailability
Drug: [14C]-GLPG3667 capsule — On Day 1, participants will receive a single oral dose of [14C]-GLPG3667
  Arms: Period 2 - Mass Balance

SUMMARY:
This is a study in healthy male volunteers to assess how a new test medicine is taken up and broken down by the body as well as its safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Male between 30 and 64 years of age (extremes included), on the date of signing the informed consent form (ICF).
* A body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.
* Has a regular daily defecation pattern (i.e. 1 to 3 times per day).
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests. Neutrophil, lymphocyte, and platelet counts must be above the lower limit of normal range. Total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be within normal range. Other clinical laboratory safety test results must be within the normal ranges or test results that are outside the normal ranges need to be considered not clinically significant in the opinion of the investigator.

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to GLPG3667 ingredients or history of a significant allergic reaction to GLPG3667 ingredients as determined by the investigator
* Treatment with any medication (including over-the-counter (OTC) and/or prescription medication, COVID-19 vaccines, dietary supplements, nutraceuticals, vitamins and/or herbal supplements), except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) in the last 2 weeks or 5 half-lives of the drug, whichever is longer, prior to the first dosing.
* Subject has participated in a [14C]-radiolabeled study within the past 12 months.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last 5 years. Occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017 (UK, 2017), cannot participate in the study.

This list only contains the key exclusion criteria.

Ages: 30 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Recovery of total radioactivity (TRA) excreted in urine expressed as a percentage of the administered dose (Ae%) | From Day 1 until at least Day 8 in Period 2
Recovery of TRA excreted in feces expressed as a percentage of the administered dose (Af%) | From Day 1 until at least Day 8 in Period 2
Recovery of TRA excreted in urine and feces expressed as a percentage of the administered dose (At%) | From Day 1 until at least Day 8 in Period 2
Percentage of TRA in plasma and excreta for metabolites of interest | From Day 1 until at least Day 8 in Period 2
Absolute oral bioavailability (F[percentage]) of GLPG3667 | From Day 1 until Day 4 in Period 1

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations. | From Day 1 through study completion, an average of 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, MD, Study Director — Galapagos NV
Locations (1):
- Quotient Sciences Limited, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No